CLINICAL TRIAL: NCT02834182
Title: Functional Magnetic Resonance Imaging Study: Theory of Mind Deficits in Schizophrenia and Bipolar Disorder
Brief Title: fMRI of Theory of Mind in Schizophrenia and Bipolar Disorder
Acronym: TOM-i
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PO16049
Record Dates: First submitted 2016-06-24; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Bipolar Disorder, Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Psychiatric Status Rating Scales; Gene Expression

ARMS (2):
- Bipolar Disorder patients and Schizophrenic patients (Experimental)
  Interventions: Behavioral: IRMf; Behavioral: Mini International Neuropsychiatric Interview; Behavioral: Positive And Negative Syndrom Scale; Behavioral: Young Mania Rating Scale; Behavioral: Hamilton Depression Scale
- Healthy Controls (Active Comparator)
  Interventions: Behavioral: IRMf; Behavioral: Mini International Neuropsychiatric Interview; Behavioral: Positive And Negative Syndrom Scale; Behavioral: Young Mania Rating Scale; Behavioral: Hamilton Depression Scale

INTERVENTIONS:
Behavioral: IRMf
Behavioral: Mini International Neuropsychiatric Interview
Behavioral: Positive And Negative Syndrom Scale
Behavioral: Young Mania Rating Scale
Behavioral: Hamilton Depression Scale

SUMMARY:
Theory of mind (TOM), a main component of social cognition processes, refers to the capacity to infer one's own and other person's mental states. Deficits in social cognition are found in patients with schizophrenia and bipolar disorder. The purpose of this study is to compare the neurofunctional profiles of schizophrenic patients, bipolar patients and healthy participants during the performance of a TOM task. Results may help to understand the neural bases of the impairments in social cognition in schizophrenia and bipolar disorder, which may in turn help to propose potential new psychosocial therapeutic approaches in these disorders.

DETAILED DESCRIPTION:
Theory of mind (TOM) refer to the cognitive ability to attribute mental states to others, which plays an essential role in social communications and interactions between individuals. In several recent papers, it was shown that TOM is impaired in schizophrenia and bipolar disorder. This impairment strongly affects the quality of life in patients suffering from these disorders. The investigators study aims to explore the neural correlates of TOM in schizophrenic and bipolar patients, in comparison with those of healthy participants. These studies will be conducted on 30 schizophrenic patients, 30 bipolar patients, and 60 healthy participants, matched on age and educational level to each patient group. The investigators expect that the study of combined behavioral (neuropsychological tests) and neuro-anatomical data will allow to understand the pathophysiology of the alteration of social cognition processes in these illnesses.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Men or women aged from 18 to 65 years-old, right-handed, with a diagnosis of bipolar -disorder or schizophrenia, according to the DSM-5 criteria
* Native French speaker
* No substantial change in treatment for 2 weeks preceding study enrollment
* Able to provide informed written and verbal consent

Healthy Controls :

* Men or women aged from 18 to 65 years-old, right-handed
* Native French speaker
* Able to provide informed written and verbal consent

Exclusion Criteria:

Patients :

* A recent alcohol and/or drug abuse or dependence (in the last six months)
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment uncorrected (visual and/or hearing)
* Contraindication to the use of MRI
* Persons under legal incapacity
* Persons who are not covered by national health insurance

Healthy Controls :

* Severe chronic psychiatric disorders including Bipolar disorder and schizophrenia
* Depression diagnostic according to DSM-5
* A personal or first-degree-relative history of bipolar disorder, schizophrenia or schizoaffective disorder according to DSM-5
* A recent alcohol and/or drug abuse or dependence (in the last six months)
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment uncorrected (visual and/or hearing)
* Contraindication to the use of MRI
* People particularly protected by the law
* Persons who are not covered by national health insurance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological test : Mini International Neuropsychiatric Interview (M.I.N.I.) | Up to 15 days after inclusion
Young Mania Rating Scale | Up to 15 days after inclusion
Hamilton Depression Scale | Up to 15 days after inclusion
Scale for the Assessment for Thought, Language and Communication | Up to 15 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Derived] Henry A, Raucher-Chene D, Obert A, Gobin P, Vucurovic K, Barriere S, Sacre S, Portefaix C, Gierski F, Caillies S, Kaladjian A. Investigation of the neural correlates of mentalizing through the Dynamic Inference Task, a new naturalistic task of social cognition. Neuroimage. 2021 Nov;243:118499. doi: 10.1016/j.neuroimage.2021.118499. Epub 2021 Aug 24. PMID 34438254